CLINICAL TRIAL: NCT04226586
Title: Nutritional Stimulation of Growth in Children With Short Stature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 239581
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2022-06

CONDITIONS: Nutritional Stunting; Growth Failure
Keywords: essential amino acids; short stature
MeSH Terms: conditions — Failure to Thrive; Dwarfism | interventions — Amino Acids, Essential; Excitatory Amino Acids; Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): * This is a double-blind study. Participants and the investigators will be blinded to the intervention.
  * Children in the treatment (intervention) arm will receive essential amino acids (EAA) twice a day.
  * Children 3 to 5 years of age will be asked to take either 8.5 g (1 serving) of EAA supplement or placebo at breakfast and at bedtime.
  * Children 6 to 11 years of age will be assigned to take either 17 g (2 servings) of EAA supplement or placebo at breakfast and at bedtime.
  * EAA and placebo dissolve easily in any liquid beverage and can be taken on empty versus full stomach.
  Interventions: Dietary Supplement: Essential Amino Acid (EAA) group
- Placebo (Placebo Comparator): * This is a double-blind study. Participants and the investigators will be blinded to the intervention.
  * Children in the placebo arm will receive placebo twice a day. EAA and placebo supplements will look and taste alike. The same flavoring ingredients (stevia blend, citric acid, malic acid, natural flavors, tartaric acid, fruit and vegetable juice for color) will be used in both products at the same amount.
  * Children 3 to 5 years of age will be asked to take either 8.5 g (1 serving) of EAA supplement or placebo at breakfast and at bedtime.
  * Children 6 to 11 years of age will be assigned to take either 17 g (2 servings) of EAA supplement or placebo at breakfast and at bedtime.
  * EAA and placebo dissolve easily in any liquid beverage and can be taken on empty versus full stomach.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Essential Amino Acid (EAA) group — Eligible children will be supplemented with Essential Amino Acids (EAA) for 6 months twice a day. Caution will be exercised to match the groups for age and sex.
  Arms: Treatment Group
Dietary Supplement: Placebo — Eligible children will be supplemented with a placebo for 6 months twice a day. Caution will be exercised to match the groups for age and sex.
  Arms: Placebo

SUMMARY:
Short stature is a frequent reason for referral to a pediatric endocrinology clinic. Short stature is especially prevalent among those with failure to thrive (whose weight is significantly below the average weight of his/her peers). The growth hormone has limited efficacy for medical treatment of short stature when the cause of short stature is not growth hormone deficiency. This study will investigate the effect of 6 months of nutritional supplement (essential amino acids) compared to placebo in the linear growth of short children who have not yet reached puberty.

ELIGIBILITY:
Inclusion Criteria:

* Ages 3 to 11 years (inclusive).
* Pre-pubertal status (i.e. Tanner stage 1 for breast development for girls and testicular enlargement for boys and pubic hair for both sexes).

Exclusion criteria:

* Ages younger than 3 years or older than 11 years.
* Medical history of a neurologic, endocrinologic, genetic, or metabolic problem known to have a direct effect on height growth. This includes, but is not limited to, children with a Growth hormone deficiency, Down syndrome, Turner syndrome, Russel-Silver syndrome, Prader-Willi syndrome, Pseudohypoparathyroidism, chronic kidney disease, malabsorptive syndromes, cancer survivors, etc.
* Currently being treated or previously treated with Growth hormone, or history of oral steroid treatment within the last 3 months.
* Being in puberty.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Linear Growth | 6 months
  Growth velocity (cm/year) will be calculated and compared between arms using the height measurements taken before and after 6 months of Essential Amino Acids vs Placebo supplementation.

SECONDARY OUTCOMES:
Body Composition | 6 months
  Lean body mass will be measured using Dual X-Ray Absorptimetry (DXA) scan and compared between arms using the measurements taken before and after 6 months of Essential Amino Acids vs Placebo supplementation.
Body Composition | 6 months
  Body fat mass will be measured using Dual X-Ray Absorptimetry (DXA) scan and compared between arms using the measurements taken before and after 6 months of Essential Amino Acids vs Placebo supplementation.
Body Composition | 6 months
  Visceral fat mass will be measured using Dual X-Ray Absorptimetry (DXA) scan and compared between arms using the measurements taken before and after 6 months of Essential Amino Acids vs Placebo supplementation.

OTHER OUTCOMES:
Serum growth factor concentrations | 6 months
  Serum concentration of Insulin-Like Growth-Factor (IGF)-I will be measured and compared between arms before and after 6 months of Essential Amino Acids vs Placebo supplementation.
Serum growth factor concentrations | 6 months
  Serum concentration of Insulin-Like Growth-Factor Binding-Protein (IGF BP)-III will be measured and compared between arms before and after 6 months of Essential Amino Acids vs Placebo supplementation.
Serum amino acid concentrations | 6 months
  Serum amino acid concentrations will be measured and compared between arms before and after 6 months of Essential Amino Acids vs Placebo supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Emir Tas, MD, Principal Investigator — Arkansas Children's Research Insitute
Locations (1):
- Emir Tas, Little Rock, Arkansas, United States